CLINICAL TRIAL: NCT03823001
Title: Evaluation of a Novel, Non-Invasive Virtual Prostate Biopsy Protocol for Patients on Active Surveillance and Patients at Risk of Harboring Low-Risk Prostate Cancer: A Prospective Non-Randomized Clinical Trial
Brief Title: Virtual Prostate Biopsy Protocol for Patients on Active Surveillance and at Risk of Prostate Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: low accrual
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CASE9818
Record Dates: First submitted 2019-01-28; First posted 2019-01-30 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Prostate Cancer
Keywords: Magnetic Resonance Imaging (MRI)
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Virtual prostate biopsy (VB) monitoring (Experimental): Prostate-specific antigen (PSA) and digital rectal exam (DRE) are standard of care for monitoring patients on active surveillance or at risk of having low-risk prostate cancer. A novel virtual biopsy (VB) monitoring protocol will be implemented:
  1. PSA bi-annually or more often according to the discretion of the urologist.
  2. Annual DRE.
  3. Visit with the urologist bi-annually.
  4. Multi-parametric MRI (mpMRI) every year for 3 years.
  5. Transrectal ultrasound (TRUS) biopsy at the end of the 3rd year.
  Interventions: Diagnostic Test: virtual biopsy (VB) monitoring protocol

INTERVENTIONS:
Diagnostic Test: virtual biopsy (VB) monitoring protocol — 1. PSA bi-annually or more often according to the discretion of the urologist.
  2. Annual DRE.
  3. Visit with the urologist bi-annually.
  4. Multi-parametric MRI (mpMRI) every year for 3 years.
  5. Transrectal ultrasound (TRUS) biopsy at the end of the 3rd year.

SUMMARY:
The purpose of this study is to examine the use of MRI surveillance for patients with no prostate cancer, potential prostate cancer, or diagnosed low-grade prostate cancer.

DETAILED DESCRIPTION:
This study will use MRI instead of prostate biopsy in combination with regularly scheduled urologist visits, interval PSA checks, and annual DRE to help establish a non-invasive method for 1) participants with a negative prostate MRI (PI-RADS 1 or 2) who have never had a biopsy; 2) participants with a positive MRI (PI-RADS score of 3, 4, or 5) and negative MRI-targeted biopsy pathology; and 3) monitoring participants with clinically diagnosed low risk prostate cancer who are on active surveillance. However, if at any point, clinical suspicion indicated either by the presence of suspicious lesions on the MRI, rising PSA, and/or positive DRE arises, then an immediate biopsy will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-naive patients with a negative prostate MRI (PI-RADS score 1 or 2); or
* Patients with a PI-RADS score of 3, 4, or 5 on MRI and a negative MR-targeted biopsy; or
* Patients on active surveillance with a negative prostate MRI (PI-RADS 1 or 2).

Exclusion Criteria:

* Positive DRE;
* PSA > 10 ng/ml or unstable PSA (doubling time <3 years) during the last year prior to enrolling in this study;
* PSAD > 0.15 (calculated using most recent PSA divided by MRI prostate volume);
* First degree relative diagnosed with prostate cancer
* First degree relative diagnosed with a BRCA2 or Lynch syndrome associated gene causing any cancer.
* Patient carries a mutation on BRCA2 or a mismatch repair gene associated with Lynch syndrome (MLHl, MSH2, MSH6, PMS2); known BRCA2 or known mismatch repair gene mutation in the family (Lynch Syndrome) and patient has not had testing; or family history consistent with BRCA2 or Lynch syndrome and there is no known BRCA2 or mismatch repair gene in the family.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Negative predictive value (NPV) of MRI (adjusted to the prostate VB protocol criteria) | Up to 3 years from start of study
  Negative predictive value (NPV) of MRI (adjusted to the prostate VB protocol criteria). This metric will determine if the the VB protocol is statistically equal to (or greater than) the negative predictive value of the standard of care TRUS prostate biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: Lee Ponsky, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the published article, after deidentification (text, tables, figures).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication
Access Criteria: To be shared with investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose.
  For individual participant data meta-analysis